CLINICAL TRIAL: NCT04834180
Title: Highest Weight Loss and Abdominal Adiposity Loss With Hypocaloric Diet Plan and Auricular Acupuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andreia Vieira (Other)
Responsible Party: Sponsor-Investigator, Andreia Vieira, Principal Investigator, Universidade do Porto
Organization: Universidade do Porto (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: uportoweightloss; uportoweightloss (Registry Identifier: uportoweightloss)
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Weight Loss; Abdominal Obesity
MeSH Terms: conditions — Weight Loss; Obesity, Abdominal | interventions — Acupuncture, Ear; Auriculotherapy; Acupressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vaccaria seeds plus diet therapy (Sham Comparator): Vaccaria seeds at the exterior side of the ear area, standard points were selected according to clinical experience in traditional Chinese medicine: Shenmen (TF4), Stomach (CO4), Hunger, Mouth (CO1), Point Zero HX1) and Sanjiao (CO17). Mustard seeds (Vaccaria ear seeds, Beijing Zhongyan Taihe Medicine, Beijing, China) were used, plus diet therapy prescribed by a licensed nutritionist.
  Interventions: Dietary Supplement: Hypocaloric diet plan; Other: Acupressure
- ASP needles plus diet therapy (Active Comparator): ASP needles on the outside of the ear standard points were selected according to clinical experience in traditional Chinese medicine: ASP gold needles, strengthening the centre with point 0 (the umbilicus) in the dominant ear, Porta Fortunae in the non-dominant ear, Barbiturate in the non-dominant ear, Psychosomatique key point in the dominant ear and the point Aggression, plus diet therapy prescribed by a licensed nutritionist.
  Interventions: Dietary Supplement: Hypocaloric diet plan; Other: Auricular Acupuncture
- only diet therapy (No Intervention): only diet therapy prescribed by a licensed nutritionist.

INTERVENTIONS:
Dietary Supplement: Hypocaloric diet plan — The hypocaloric diet is one in which there is a reduction of daily calories or foods with high caloric density usually in order to aid weight loss.
  Arms: ASP needles plus diet therapy; Vaccaria seeds plus diet therapy
Other: Auricular Acupuncture — Auriculotherapy is a technique derived from traditional acupuncture developed into a distinct treatment system of its own. It is based on either, the introduction of needles (auricular acupuncture), or pressure with Vaccaria seeds (acupressure). Those forms of auriculotherapy are applied on a set of anatomical maps at a specific point in the auricular region.
  Other Names: Auriculotherapy
  Arms: ASP needles plus diet therapy
Other: Acupressure — Auriculotherapy is a technique derived from traditional acupuncture developed into a distinct treatment system of its own. It is based on either, the introduction of needles (auricular acupuncture), or pressure with Vaccaria seeds (acupressure). Those forms of auriculotherapy are applied on a set of anatomical maps at a specific point in the auricular region.
  Other Names: Auriculotherapy
  Arms: Vaccaria seeds plus diet therapy

SUMMARY:
The implications of obesity, especially visceral fat, in health are well known. It would be desirable to control obesity by safe and effective treatment modalities. Aim: To assess the effectiveness of Auricular Acupuncture (AA) on body weight loss in a Portuguese sample.

DETAILED DESCRIPTION:
Methods: After a pre-study, a prospective experimental randomized, controlled and single-blinded study was conducted. The sample included 31 adult women with ages ranging from 20 to 51 years old. The groups had a frequency of physical activity ≥ 2 and ≤ 4 times per week. Individuals with BMI ≤ 24.9 Kg/m2 and pregnant women excluded from the study. All participants were then randomized into one of three groups: group 1 was treated with Vaccaria seeds plus diet therapy, group 2 with ASP needles plus diet therapy and finally, group 3 received only diet therapy. A licensed nutritionist prescribed the hypocaloric diet plan. Baseline evaluation included anthropometric measures collected according to standardized procedures. They received two treatments per week for a total of 6 weeks. After one month of follow-up, all the anthropometric measures were reevaluated. Main Parameters: Weight/body composition by bioelectrical impedance analysis. Secondary parameters: Waist to height ratio (WHtR), weight and Body Mass Index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Unfamiliar to acupuncture

Exclusion Criteria:

* Psychotropic medication
* Psychiatric or thyroid disorders
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — adults
Enrollment: 31 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-12-15 (Actual)

PRIMARY OUTCOMES:
Weight (kg) | 1 month
  TANITA® bio-impedance scale (model 762)
Waist Perimeter (cm) | 1 month
  tape measure from SECA® (model 203)
height (cm) | 1 month
  SECA® stadiometer (model 208)
body fat (%) | 1 month
  TANITA® bio-impedance scale (model 762)
Body mass index (kg/m2) | 1 month
  Body mass index is defined as the body mass divided by the square of the body height.
Waist-to-height ratio (cm2) | 1 month
  The WHTR was obtained by dividing the waist circumference (cm) by height (cm).

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR